CLINICAL TRIAL: NCT03442725
Title: A Phase I, Open-label Study to Compare the Pharmacokinetics of Telotristat Ethyl and Its Metabolite in Subjects With Impaired Renal Function to Healthy Subjects With Normal Renal Function After a Single Dose of Telotristat Etiprate
Brief Title: Study to Compare a Dose of Telotristat Etiprate in Subjects With Renal Impairment With Matched Subjects With Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D-FR-01017-002; 2017-003948-20 (EudraCT Number)
Record Dates: First submitted 2018-01-26; First posted 2018-02-22 (Actual); Results first posted 2019-09-13 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-03

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — telotristat; telotristat ethyl

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Severely decreased renal function group (Experimental): Subjects will receive a single oral 250-mg tablet dose of Telotristat etiprate (Xermelo® 250 mg) on day 1 under fed conditions (i.e. between 15 minutes before and 1 hour after the meal or snack).
  Interventions: Drug: Telotristat etiprate
- Normal renal function group (Active Comparator): Subjects will receive a single oral 250-mg tablet dose of Telotristat etiprate (Xermelo® 250 mg) on day 1 under fed conditions (i.e. between 15 minutes before and 1 hour after the meal or snack).
  Interventions: Drug: Telotristat etiprate
- Mildly decreased renal function group (Experimental): Subjects will receive a single oral 250-mg tablet dose of Telotristat etiprate (Xermelo® 250 mg) on day 1 under fed conditions (i.e. between 15 minutes before and 1 hour after the meal or snack).
  Interventions: Drug: Telotristat etiprate
- Moderately decreased renal function group (Experimental): Subjects will receive a single oral 250-mg tablet dose of Telotristat etiprate (Xermelo® 250 mg) on day 1 under fed conditions (i.e. between 15 minutes before and 1 hour after the meal or snack).
  Interventions: Drug: Telotristat etiprate

INTERVENTIONS:
Drug: Telotristat etiprate — Oral administration of 1 tablet of Xermelo® containing telotristat etiprate equivalent to 250 mg telotristat ethyl.
  Other Names: Xermelo®

SUMMARY:
Renal excretion is a minor elimination route of telotristat etiprate. So this trial is intended to assess the drug behaviour in subjects with decreased renal function.

This is a staged study with Part B contingent upon the results of Part A. Part A will enrol a total of 16 subjects, eight with severely impaired renal function and eight healthy subjects. Part B with enrol a total of 16 subjects, eight subjects in each additional renal function group, i.e. mildly impaired renal function group and moderately impaired group.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* Provision of written informed consent prior to any study related procedure.
* Men and women enrolling in the study must be at least 18 years of age at the time of giving informed consent.
* Women of childbearing potential must agree to use an adequate double-barrier method of contraception during the study and for 30 days after discharge.
* Men must agree to use an adequate, double barrier method of contraception during the study and for 30 days after discharge.

Additionally, for subjects with renal impaired function:

* Clinical diagnosis of renal impaired function that has been stable for more than 3 months prior to dosing
* Renal impaired function classified as mild, moderate, or severe.
* Under stable medication regimen, i.e. not starting new therapy(ies) or significant changing dosage(s) within at least 1 month prior to dosing, as determined by the investigator.
* Stable and appropriately managed relative to chronic diseases (e.g. diabetes, hypertension) as determined by medical history, physical examination, ECGs, and clinical laboratory tests.

Additionally, for healthy subjects with normal renal function:

* Each subject will be demographically-matched to one of the subjects with severely impaired renal function for gender, age (± 10 years), BMI (± 20%).
* Clinical laboratory test results must be strictly within the normal laboratory reference ranges for urea, creatinine, protein, and albumin.

Exclusion Criteria:

All subjects:

* Existence of any surgical or medical condition that, in the judgment of the investigator, might interfere with the absorption, distribution, metabolism, or excretion of telotristat etiprate (including bariatric surgery, or any other gastrointestinal surgery, excepting appendectomy and hernia repair, which are acceptable).
* History of any major surgery within six months or anticipated surgery prior to Day-1.
* Patients with hereditary problems of galactose intolerance (lactase deficiency or glucose-galactose malabsorption).
* History of any active infection within 30 days prior to Day-1, if deemed clinically significant by the investigator.
* Positive hepatitis panel results (including hepatitis B surface antigen and hepatitis virus C ribonucleic acid).
* Positive results for human immunodeficiency virus, or who has received diagnosis for acquired immunodeficiency syndrome.
* Positive urine screen for drugs of abuse (not including cotinine).
* Consumption of alcohol within 48 hours prior to Day-1 (as confirmed by alcohol breath screen) and for the duration of the confinement period.
* Smoking more than ten cigarettes per day or equivalent; unable or unwilling to refrain from smoking and tobacco use for two hours prior to dosing and four hours after dose administration.
* Consumption of caffeine- and/or xanthine-containing products (e.g. cola, coffee, tea, chocolate) on Day-1 until 24 hours postdose.
* Consumption of grapefruit, Seville oranges, and grapefruit- or Seville orange-containing products within 72 hours prior to Day-1 and for the duration of the confinement period.
* Use of any medication (prescription or over-the-counter), Chinese herbal medications or herbal tea, energy drinks, herbal products (e.g. St. John's wort, garlic), or supplements/supra therapeutic doses of vitamins within 14 days prior to Day-1 and up to Day 4 after dosing, apart from those approved by the investigator.
* Women who are breastfeeding or are planning to become pregnant during the study.

Additionally, for renal impaired subjects:

* Clinically significant physical (e.g. oedema in heavy subjects with renal impaired function), laboratory, or ECG findings (apart from those parameters which are related to impaired renal function or underlying disease e.g. diabetes, hypertension) that, in the opinion of the investigator, may interfere with any aspect of the study conduct or interpretation of the results.
* Glycated haemoglobin A1c ≥ 9%.

Additionally, for healthy subjects with normal renal function:

* Clinically significant illness or disease including cardiac, pulmonary, hepato-biliary, gastrointestinal, or endocrinology, or cancer within the last 5 years (except localised or in situ non-melanoma skin cancer), as determined by medical history, physical examination, laboratory tests, and 12-lead ECGs.
* Clinically significant physical, laboratory, or ECG findings that, in the opinion of the investigator, may interfere with any aspect of the study conduct or interpretation of the results.
* History of renal disease.
* History of alcohol or drug abuse within 2 years prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (4):
- A.T.C. s.a., Clinical Pharmacology Unit, CHU Sart-Tilman, Liège, Belgium
- CRS Clinical Research Services Kiel GmbH, Kiel, Germany
- ARENSIA Exploratory Medicine Phase I Unit, Republican Clinical Hospital, Chisinau, Moldova
- ARENSIA Unit in Spitalul de Nefrologie, Bucharest, Romania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 16 subjects were recruited in this open label, single dose study between February and May 2018. Recruited subjects were split evenly between 2 groups (control group and test group).
Pre-assignment Details: The control group comprised 8 healthy subjects with normal renal function and who were demographically matched to test group by age (±10 years), sex and body mass index (BMI) (±20%). 8 subjects with severely impaired renal function but not requiring dialysis were recruited into the test group.
Groups:
- Healthy Subjects (Control Group): Subjects with normal renal function (estimated glomerular filtration rate [eGFR] ≥90 millilitres/minute/1.73 metres squared [mL/min/1.73 m²]) received a single oral dose of 250 milligrams (mg) telotristat etiprate given under fed conditions (between 15 minutes before and 1 hour after the meal or snack) on Day 1.
- Severe Renal Impairment (Test Group): Subjects with severely decreased renal function (eGFR <30 mL/min/1.73 m², not requiring dialysis) received a single oral dose of 250 mg telotristat etiprate given under fed conditions (between 15 minutes before and 1 hour after the meal or snack) on Day 1.
Period: Overall Study
Arm/Group | Healthy Subjects (Control Group) | Severe Renal Impairment (Test Group)
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Subjects (Control Group): Subjects with normal renal function (eGFR ≥90 mL/min/1.73 m²) received a single oral dose of 250 mg telotristat etiprate given under fed conditions (between 15 minutes before and 1 hour after the meal or snack) on Day 1.
- Total: Total of all reporting groups
Arm/Group | Healthy Subjects (Control Group) | Severe Renal Impairment (Test Group) | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Romania | 3 | 3 | 6
  Belgium | 1 | 3 | 4
  Moldova | 2 | 0 | 2
  Germany | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Total Telotristat Ethyl, LP-778902 and LP-951757
Description: Blood samples were collected to determine plasma levels of telotristat ethyl, its active metabolite LP-778902 (also known as telotristat) and the inactive metabolite LP-951757 using a validated, specific and sensitive liquid chromatography-tandem mass spectrometry (LC-MS/MS) bioanalytical method with a lower limit of quantitation (LOQ) of 0.5 nanograms (ng)/mL for telotristat ethyl and 2 ng/mL for LP-778902 and LP-951757.
  Cmax was determined using non-compartmental analysis.
Time Frame: Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours), Day 2 (24 hours), Day 3 (48 hours) and Day 4 (72 hours)
Population: The pharmacokinetic (PK) population included all subjects who received the single oral dose of study drug and had no major protocol deviations affecting the PK variables and for whom the renal function group was assessable and who had a sufficient number of plasma concentrations to estimate the main PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Healthy Subjects (Control Group) | Severe Renal Impairment (Test Group)
Number analyzed (Participants) | 8 | 8
ng/mL
  Telotristat Ethyl | 3.81 (98.9) | 4.94 (116)
  LP-778902 | 533 (58.1) | 759 (52.9)
  LP-951757 | 65.2 (46.0) | 45.6 (80.2)
Statistical Analysis 1: Comparison: Healthy Subjects (Control Group) vs Severe Renal Impairment (Test Group); Analysis of variance (ANOVA) comparison of Cmax for telotristat ethyl between test group versus the control group; Test type: Other; Geometric Mean Ratio = 1.297, 90% CI 2-sided [0.600 to 2.805]
Statistical Analysis 2: Comparison: Healthy Subjects (Control Group) vs Severe Renal Impairment (Test Group); ANOVA comparison of Cmax for LP-778902 between test group versus the control group; Test type: Other; Geometric Mean Ratio = 1.423, 90% CI 2-sided [0.901 to 2.247]

2. Primary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Total Telotristat Ethyl, LP-778902 and LP-951757
Description: Blood samples were collected to determine plasma levels of telotristat ethyl, its active metabolite LP-778902 (also known as telotristat) and the inactive metabolite LP-951757 using a validated, specific and sensitive LC-MS/MS bioanalytical method with a LOQ of 0.5 ng/mL for telotristat ethyl and 2 ng/mL for LP-778902 and LP-951757.
  Tmax was determined using non-compartmental analysis.
Time Frame: Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours), Day 2 (24 hours), Day 3 (48 hours) and Day 4 (72 hours)
Population: The PK population included all subjects who received the single oral dose of study drug and had no major protocol deviations affecting the PK variables and for whom the renal function group was assessable and who had a sufficient number of plasma concentrations to estimate the main PK parameters.
Measure: Median (Full Range); unit: hours
Arm/Group | Healthy Subjects (Control Group) | Severe Renal Impairment (Test Group)
Number analyzed (Participants) | 8 | 8
hours
  Telotristat Ethyl | 1.03 [0.500 to 3.00] | 1.00 [0.500 to 3.00]
  LP-778902 | 2.00 [1.00 to 4.00] | 2.50 [1.00 to 3.00]
  LP-951757 | 4.00 [3.00 to 8.00] | 4.00 [2.02 to 6.00]
Statistical Analysis 1: Comparison: Healthy Subjects (Control Group) vs Severe Renal Impairment (Test Group); Comparison of tmax for telotristat ethyl between test group versus the control group; Test type: Other — Estimate of the median difference and 90% confidence intervals (CIs) was determined by Hodges-Lehmann estimation; p = 0.7452, Wilcoxon (Mann-Whitney); Median Difference = 0.000, 90% CI 2-sided [-1.000 to 0.950]
Statistical Analysis 2: Comparison: Healthy Subjects (Control Group) vs Severe Renal Impairment (Test Group); Comparison of tmax for LP-778902 between test group versus the control group; Test type: Other — Estimate of the median difference and 90% CIs was determined by Hodges-Lehmann estimation; p = 0.7039, Wilcoxon (Mann-Whitney); Median Difference = 0.000, 90% CI 2-sided [-1.000 to 1.000]

3. Primary Outcome: Apparent Terminal Elimination Half-Life (t1/2) of Total Telotristat Ethyl, LP-778902 and LP-951757
Description: Blood samples were collected to determine plasma levels of telotristat ethyl, its active metabolite LP-778902 (also known as telotristat) and the inactive metabolite LP-951757 using a validated, specific and sensitive LC-MS/MS bioanalytical method with a LOQ of 0.5 ng/mL for telotristat ethyl and 2 ng/mL for LP-778902 and LP-951757.
  T1/2 was determined using non-compartmental analysis.
Time Frame: Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours), Day 2 (24 hours), Day 3 (48 hours) and Day 4 (72 hours)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Healthy Subjects (Control Group) | Severe Renal Impairment (Test Group)
Number analyzed (Participants) | 8 | 8
hours
  Telotristat Ethyl: number analyzed (Participants) | 4 | 4
  Telotristat Ethyl | NA (NA) — Result was not calculated when more than one-third of the values were below the limit of quantification (BLQ) at a single time point. | NA (NA) — Result was not calculated when more than one-third of the values were BLQ at a single time point.
  LP-778902 | 9.05 (3.02) | 8.31 (1.51)
  LP-951757: number analyzed (Participants) | 7 | 5
  LP-951757 | 11.5 (4.65) | 9.93 (4.45)

4. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity (AUC0-inf) of Total Telotristat Ethyl, LP-778902 and LP-951757
Description: Blood samples were collected to determine plasma levels of telotristat ethyl, its active metabolite LP-778902 (also known as telotristat) and the inactive metabolite LP-951757 using a validated, specific and sensitive LC-MS/MS bioanalytical method with a LOQ of 0.5 ng/mL for telotristat ethyl and 2 ng/mL for LP-778902 and LP-951757.
  AUC0-inf was determined using non-compartmental analysis.
Time Frame: Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours), Day 2 (24 hours), Day 3 (48 hours) and Day 4 (72 hours)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | Healthy Subjects (Control Group) | Severe Renal Impairment (Test Group)
Number analyzed (Participants) | 8 | 8
ng*hour/mL
  Telotristat Ethyl: number analyzed (Participants) | 1 | 2
  Telotristat Ethyl | NA (NA) — Result was not calculated when more than one-third of the values were BLQ at a single time point. | NA (NA) — Result was not calculated when more than one-third of the values were BLQ at a single time point.
  LP-778902 | 1652 (42.7) | 2488 (77.9)
  LP-951757: number analyzed (Participants) | 7 | 5
  LP-951757 | 876 (66.0) | 511 (115)
Statistical Analysis 1: Comparison: Healthy Subjects (Control Group) vs Severe Renal Impairment (Test Group); ANOVA comparison of AUC0-inf for LP-778902 between test group versus the control group; Test type: Other; Geometric Mean Ratio = 1.506, 90% CI 2-sided [0.914 to 2.480]

5. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to Time Corresponding to the Last Quantifiable Concentration (AUC0-tlast) of Total Telotristat Ethyl, LP-778902 and LP-951757
Description: Blood samples were collected to determine plasma levels of telotristat ethyl, its active metabolite LP-778902 (also known as telotristat) and the inactive metabolite LP-951757 using a validated, specific and sensitive LC-MS/MS bioanalytical method with a LOQ of 0.5 ng/mL for telotristat ethyl and 2 ng/mL for LP-778902 and LP-951757.
  AUC0-tlast was determined using non-compartmental analysis.
Time Frame: Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours), Day 2 (24 hours), Day 3 (48 hours) and Day 4 (72 hours)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | Healthy Subjects (Control Group) | Severe Renal Impairment (Test Group)
Number analyzed (Participants) | 8 | 8
ng*hour/mL
  Telotristat Ethyl: number analyzed (Participants) | 1 | 2
  Telotristat Ethyl | NA (NA) — Result was not calculated when more than one-third of the values were BLQ at a single time point. | NA (NA) — Result was not calculated when more than one-third of the values were BLQ at a single time point.
  LP-778902 | 1637 (43.3) | 2475 (78.3)
  LP-951757: number analyzed (Participants) | 7 | 5
  LP-951757 | 845 (64.4) | 494 (118)
Statistical Analysis 1: Comparison: Healthy Subjects (Control Group) vs Severe Renal Impairment (Test Group); ANOVA comparison of AUC0-tlast for LP-778902 between test group versus the control group; Test type: Other; Geometric Mean Ratio = 1.512, 90% CI 2-sided [0.915 to 2.498]

6. Primary Outcome: Apparent First Order Terminal Elimination Rate Constant (λz) of Total Telotristat Ethyl, LP-778902 and LP-951757
Description: Blood samples were collected to determine plasma levels of telotristat ethyl, its active metabolite LP-778902 (also known as telotristat) and the inactive metabolite LP-951757 using a validated, specific and sensitive LC-MS/MS bioanalytical method with a LOQ of 0.5 ng/mL for telotristat ethyl and 2 ng/mL for LP-778902 and LP-951757.
  λz was determined using non-compartmental analysis.
Time Frame: Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours), Day 2 (24 hours), Day 3 (48 hours) and Day 4 (72 hours)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour^-1
Arm/Group | Healthy Subjects (Control Group) | Severe Renal Impairment (Test Group)
Number analyzed (Participants) | 8 | 8
hour^-1
  Telotristat Ethyl: number analyzed (Participants) | 4 | 4
  Telotristat Ethyl | NA (NA) — Result was not calculated when more than one-third of the values were BLQ at a single time point. | NA (NA) — Result was not calculated when more than one-third of the values were BLQ at a single time point.
  LP-778902 | 0.0890 (0.0469) | 0.0871 (0.0236)
  LP-951757: number analyzed (Participants) | 7 | 5
  LP-951757 | 0.0686 (0.0238) | 0.0821 (0.0381)

7. Primary Outcome: Apparent Total Clearance From Plasma (CL/F) of Total Telotristat Ethyl
Description: Blood samples were collected to determine plasma levels of telotristat ethyl using a validated, specific and sensitive LC-MS/MS bioanalytical method with a LOQ of 0.5 ng/mL.
  CL/F was determined using non-compartmental analysis.
Time Frame: Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours), Day 2 (24 hours), Day 3 (48 hours) and Day 4 (72 hours)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Litres/hour
Arm/Group | Healthy Subjects (Control Group) | Severe Renal Impairment (Test Group)
Number analyzed (Participants) | 1 | 2
Litres/hour | NA (NA) — Result was not calculated when more than one-third of the values were BLQ at a single time point. | NA (NA) — Result was not calculated when more than one-third of the values were BLQ at a single time point.

8. Primary Outcome: Apparent Volume of Distribution (Vd/F) of Total Telotristat Ethyl
Description: Blood samples were collected to determine plasma levels of telotristat ethyl using a validated, specific and sensitive LC-MS/MS bioanalytical method with a LOQ of 0.5 ng/mL.
  Vd/F was determined using non-compartmental analysis.
Time Frame: Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours), Day 2 (24 hours), Day 3 (48 hours) and Day 4 (72 hours)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Healthy Subjects (Control Group) | Severe Renal Impairment (Test Group)
Number analyzed (Participants) | 1 | 2
Litres | NA (NA) — Result was not calculated when more than one-third of the values were BLQ at a single time point. | NA (NA) — Result was not calculated when more than one-third of the values were BLQ at a single time point.

9. Primary Outcome: Percentage of Unbound Plasma Fraction (fu) of Total Telotristat Ethyl, LP-778902 and LP-951757
Description: Plasma protein binding was assessed using equilibrium dialysis followed by LC-MS/MS for determination of unbound drug concentrations. The plasma protein binding of telotristat ethyl, LP-778902 and LP-951757 was assessed and the percentage of fu was calculated as the mean over time of the mean of the available replicates.
Time Frame: Day 1 (0.5, 1, 2 and 3 hours post-dose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of fu
Arm/Group | Healthy Subjects (Control Group) | Severe Renal Impairment (Test Group)
Number analyzed (Participants) | 8 | 8
Percentage of fu
  Telotristat Ethyl | NA (NA) — Not determined as only 1 subject displayed a value above the LOQ. | NA (NA) — Not determined as only 1 subject displayed a value above the LOQ.
  LP-778902 | 0.115 (0.0589) | 0.134 (0.0524)
  LP-951757 | 0.135 (0.295) | 0.0608 (0.0923)
Statistical Analysis 1: Comparison: Healthy Subjects (Control Group) vs Severe Renal Impairment (Test Group); ANOVA comparison of fu of LP-778902 between test group versus the control group; Test type: Other; Arithmetic Mean Difference = 0.019, 90% CI 2-sided [-0.030 to 0.068]

10. Primary Outcome: Cmax for the Unbound Fraction (Cmaxu) of Unbound Telotristat Ethyl, LP-778902 and LP-951757
Description: Cmaxu of unbound telotristat ethyl and its active metabolite LP-778902 (also known as telotristat) and the inactive metabolite LP-951757 was calculated using the unbound fraction fu (defined for each subject as the mean over all time points of the mean of fu) and determined using non-compartmental analysis.
Time Frame: Day 1 (0.5, 1, 2 and 3 hours post-dose)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Healthy Subjects (Control Group) | Severe Renal Impairment (Test Group)
Number analyzed (Participants) | 8 | 8
ng/mL
  Telotristat Ethyl | NA (NA) — Not determined as only 1 subject displayed an unbound fraction value above the LOQ. | NA (NA) — Not determined as only 1 subject displayed an unbound fraction value above the LOQ.
  LP-778902 | 0.554 (113) | 0.957 (70.7)
  LP-951757 | 0.0528 (215) | 0.0779 (84.0)
Statistical Analysis 1: Comparison: Healthy Subjects (Control Group) vs Severe Renal Impairment (Test Group); ANOVA comparison of Cmaxu for LP-778902 between test group versus the control group; Test type: Other; Geometric Mean Ratio = 1.727, 90% CI 2-sided [0.866 to 3.443]

11. Primary Outcome: AUC0-inf for the Unbound Fraction (AUC0-infu) of Unbound Telotristat Ethyl, LP-778902 and LP-951757
Description: AUC0-infu of unbound telotristat ethyl and its active metabolite LP-778902 (also known as telotristat) and the inactive metabolite LP-951757 was calculated using the unbound fraction fu (defined for each subject as the mean over all time points of the mean of fu) and determined using non-compartmental analysis.
Time Frame: Day 1 (0.5, 1, 2 and 3 hours post-dose)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | Healthy Subjects (Control Group) | Severe Renal Impairment (Test Group)
Number analyzed (Participants) | 8 | 8
ng*hour/mL
  Telotristat Ethyl: number analyzed (Participants) | 1 | 2
  Telotristat Ethyl | NA (NA) — Result was not calculated when more than one-third of the values were BLQ at a single time point. | NA (NA) — Result was not calculated when more than one-third of the values were BLQ at a single time point.
  LP-778902 | 1.72 (90.3) | 3.14 (99.2)
  LP-951757: number analyzed (Participants) | 7 | 5
  LP-951757 | 0.955 (237) | 1.06 (NA) — Not determined due to insufficient values different from 0.
Statistical Analysis 1: Comparison: Healthy Subjects (Control Group) vs Severe Renal Impairment (Test Group); ANOVA comparison of AUC0-infu for LP-778902 between test group versus the control group; Test type: Other; Geometric Mean Ratio = 1.828, 90% CI 2-sided [0.903 to 3.699]

12. Primary Outcome: AUC0-tlast for the Unbound Fraction (AUC0-tlastu) of Unbound Telotristat Ethyl, LP-778902 and LP-951757
Description: AUC0-tlastu of unbound telotristat ethyl and its active metabolite LP-778902 (also known as telotristat) and the inactive metabolite LP-951757 was calculated using the unbound fraction fu (defined for each subject as the mean over all time points of the mean of fu) and determined using non-compartmental analysis.
Time Frame: Day 1 (0.5, 1, 2 and 3 hours post-dose)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | Healthy Subjects (Control Group) | Severe Renal Impairment (Test Group)
Number analyzed (Participants) | 8 | 8
ng*hour/mL
  Telotristat Ethyl: number analyzed (Participants) | 1 | 2
  Telotristat Ethyl | NA (NA) — Result was not calculated when more than one-third of the values were BLQ at a single time point. | NA (NA) — Result was not calculated when more than one-third of the values were BLQ at a single time point.
  LP-778902 | 1.70 (91.2) | 3.12 (99.6)
  LP-951757: number analyzed (Participants) | 7 | 5
  LP-951757 | 0.928 (234) | 1.05 (NA) — Not determined due to insufficient values different from 0.
Statistical Analysis 1: Comparison: Healthy Subjects (Control Group) vs Severe Renal Impairment (Test Group); ANOVA comparison of AUC0-tlastu for LP-778902 between test group versus the control group; Test type: Other; Geometric Mean Ratio = 1.835, 90% CI 2-sided [0.904 to 3.726]

13. Primary Outcome: Metabolic Ratios (MR) of Cmax (LP-778902/Telotristat Ethyl)
Description: The following MRs of Cmax were calculated:
  MRCmax = (Cmax LP-778902)/(Cmax telotristat ethyl)
  MRCmaxTotal = (Cmax LP-778902)/(Cmax LP-778902+Cmax telotristat ethyl)
  The ratios were also normalised by molecular weight (MW) of the metabolites (telotristat ethyl: MW=575 grams/mole (g/mol) and LP-778902: MW=547 g/mol). Both the normalised and not normalised ratios are presented.
Time Frame: Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours), Day 2 (24 hours), Day 3 (48 hours) and Day 4 (72 hours)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Healthy Subjects (Control Group) | Severe Renal Impairment (Test Group)
Number analyzed (Participants) | 8 | 8
Ratio
  MRCmax - not normalised | 154 (68.9) | 204 (143)
  MRCmax - normalised | 162 (72.4) | 215 (151)
  MRCmaxTotal - not normalised | 0.992 (0.00410) | 0.991 (0.00996)
  MRCmaxTotal - normalised | 0.993 (0.00391) | 0.991 (0.00949)

14. Secondary Outcome: Amount of Unchanged Telotristat Ethyl and LP-778902 Excreted in Urine.
Description: For assessment of urine PK parameters, the amount of unchanged telotristat ethyl and its active metabolite LP-778902 (also known as telotristat) excreted in urine was determined.
Time Frame: Day 1 (predose and 0 to 4 hours, 4 to 8 hours, 8 to 12 hours, 12 to 24 hours post-dose), Day 2 (24 to 48 hours post-dose), Day 3 (48 to 72 hours post-dose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | Healthy Subjects (Control Group) | Severe Renal Impairment (Test Group)
Number analyzed (Participants) | 8 | 8
ng
  Telotristat Ethyl: All timepoints: number analyzed (Participants) | 0 | 0
  LP-778902: Pre-dose | 0 (0) | 0 (0)
  LP-778902: 0-4 hours post-dose | 88966 (50003) | 19293 (9447)
  LP-778902: 4-8 hours post-dose | 152419 (48649) | 42976 (22836)
  LP-778902: 8-12 hours post-dose | 173416 (49499) | 47955 (25522)
  LP-778902: 12-24 hours post-dose | 185970 (47726) | 51970 (27925)
  LP-778902: 24-48 hours post-dose | 191999 (48110) | 53997 (29262)
  LP-778902: 48-72 hours post-dose | 193880 (48123) | 54397 (29546)

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were recorded from Day 1 to the end of study visit between Day 8 and Day 15 (overall timeframe: up to 15 days).
Groups:
- Healthy Subjects (Control Group): Subjects with normal renal function (eGFR ≥90 mL/min/1.73 m²) received a single dose of 250 mg telotristat etiprate given under fed conditions (between 15 minutes before and 1 hour after the meal or snack) on Day 1.
- Severe Renal Impairment (Test Group): Subjects with severely decreased renal function (eGFR <30 mL/min/1.73 m², not requiring dialysis) received a single dose of 250 mg telotristat etiprate given under fed conditions (between 15 minutes before and 1 hour after the meal or snack) on Day 1.
Arm/Group | Healthy Subjects (Control Group) | Severe Renal Impairment (Test Group)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Subjects (Control Group) (N=8) | Severe Renal Impairment (Test Group) (N=8)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Monocyte count increased (Investigations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (2)

LIMITATIONS AND CAVEATS:
In accordance with the statistical analysis plan, PK parameters were not calculated if more than one-third of the values were BLQ at a single time point. No statistical comparisons were performed on PK parameters for LP-951757.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/25/NCT03442725/SAP_000.pdf
  • Study Protocol (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT03442725/Prot_001.pdf